CLINICAL TRIAL: NCT00462215
Title: An Open Label Phase III Study of a Vero Cell-Derived Whole Virus H5N1 Influenza Vaccine to Assess the Immunogenicity and Safety and to Investigate the Need for and Timing of a Booster Vaccination
Brief Title: Phase 3 Immunogenicity and Safety Study of an Inactivated H5N1 Influenza Vaccine (Whole Virion, Vero Cell Derived)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Esther-Maria Imre, Clinical Project Manager, Baxter Healthcare Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 810601
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2010-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 6-month booster vaccination with the H5N1 vaccine containing 3.75 mg HA antigen strain A/Vietnam/1203/2004
  Interventions: Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen
- 2 (Experimental): Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 6-month booster vaccination with the H5N1 vaccine containing 7.5 mg HA antigen strain A/Vietnam/1203/2004
  Interventions: Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen
- 3 (Experimental): Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 6-month booster vaccination with the H5N1 vaccine containing 3.75 mg HA antigen strain A/Indonesia/05/2005
  Interventions: Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen
- 4 (Experimental): Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 6-month booster vaccination with the H5N1 vaccine containing 7.5 mg HA antigen strain A/Indonesia/05/2005
  Interventions: Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen
- 5 (Experimental): Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 12-month booster vaccination with the H5N1 vaccine containing 3.75 mg HA antigen of the A/Indonesia/05/2005 strain
  Interventions: Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen
- 6 (Experimental): Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 24-month booster vaccination with the H5N1 vaccine containing 3.75 mg HA antigen of the A/Indonesia/05/2005 strain
  Interventions: Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen

INTERVENTIONS:
Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen — Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 6-month booster vaccination with the H5N1 vaccine containing 3.75 mg HA antigen strain A/Vietnam/1203/2004
  Arms: 1
Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen — Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 6-month booster vaccination with the H5N1 vaccine containing 7.5 mg HA antigen strain A/Vietnam/1203/2004
  Arms: 2
Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen — Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 6-month booster vaccination with the H5N1 vaccine containing 3.75 mg HA antigen strain A/Indonesia/05/2005
  Arms: 3
Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen — Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 6-month booster vaccination with the H5N1 vaccine containing 7.5 mg HA antigen strain A/Indonesia/05/2005
  Arms: 4
Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen — Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 12-month booster vaccination with the H5N1 vaccine containing 3.75 mg HA antigen of the A/Indonesia/05/2005 strain
  Arms: 5
Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen — Vaccination on Day 0 and Day 21 with the whole virion, Vero cell-derived influenza vaccine containing 7.5 µg H5N1 hemagglutinin (HA) antigen (without adjuvant) of the A/Vietnam/1203/2004 strain + 24-month booster vaccination with the H5N1 vaccine containing 3.75 mg HA antigen of the A/Indonesia/05/2005 strain
  Arms: 6

SUMMARY:
The objectives of this study are to assess the immune response as well as the safety and tolerability of an H5N1 influenza vaccine in an adult and elderly population. Further, the study will assess the need for a booster vaccination and whether a 6-month booster or a 12-month booster is more appropriate. An independent data safety monitoring board will review and evaluate the safety data obtained in this study on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects will be eligible for participation in this study if they:

* Are 18 to 59 years of age on the day of screening (for Stratum A only),
* Are 60 years of age and older on the day of screening (for Stratum B only),
* Have an understanding of the study, agree to its provisions, and give written informed consent prior to study entry,
* Are clinically healthy (in a physical condition such that the physician would have no reservations vaccinating with an influenza vaccine outside the scope of a clinical study),
* Agree to keep a daily record of symptoms,
* If female and capable of bearing children - have a negative urine pregnancy test result at study entry and agree to employ adequate birth control measures for the duration of the study.

Exclusion Criteria:

Subjects will be excluded from participation in this study if they:

* Have a history of exposure to H5N1 virus or a history of vaccination with an H5N1 influenza vaccine,
* Are at high risk of contracting H5N1 influenza infection (e.g. poultry workers),
* Suffer from or have a history of a significant cardiovascular, pulmonary, neurological, hepatic, rheumatic, autoimmune, hematological, metabolic or renal disorder,
* Are unable to lead an independent life as a result of either physical or mental handicap,
* Suffer from any kind of immunodeficiency,
* Suffer from a disease or were undergoing a treatment within 30 days prior to study entry or are currently undergoing a form of treatment that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (>800µg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs,
* Have a history of severe allergic reactions or anaphylaxis,
* Have a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating,
* Have received a blood transfusion or immunoglobulins within 90 days of study entry,
* Have donated blood or plasma within 30 days of study entry,
* Have received any live vaccine within 4 weeks or inactivated vaccine within 2 weeks prior to vaccination in this study,
* Have a functional or surgical asplenia,
* Have a known or suspected problem with alcohol or drug abuse,
* Were administered an investigational drug within six weeks prior to study entry or are concurrently participating in a clinical study that includes the administration of an investigational product,
* Are a member of the team conducting this study or are in a dependent relationship with the study investigator. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator,
* If female, are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-06 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with antibody response to the vaccine strain (A/Vietnam/1203/2004) associated with protection 21 days after the second vaccination defined as titer measured by microneutralization (MN) test >= 20. | 21 days after the second vaccination (= Day 42 in the study)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, MD, Principal Investigator — Baxter Healthcare Corporation
Locations (2):
- University Hospital, Department of Clinical Pharmacology, General Hospital Vienna, Vienna, Austria
- University Hospital Mainz, Mainz, Germany